CLINICAL TRIAL: NCT04341129
Title: Abbreviated MRI Protocol: Initial Experience With Dotarem® (Gadoterate Meglumine)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB19-2074; I002672 (Other Grant/Funding Number: Guerbet)
Record Dates: First submitted 2020-03-26; First posted 2020-04-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms; Breast Diseases; Breast Fibroadenoma; Breast Cancer
Keywords: Breast; Breast Cancer; Invasive Ductal Cancer; Ductal Carcinoma in situ; Breast Neoplasm; Fibroadenoma
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases; Fibroadenoma; Carcinoma, Intraductal, Noninfiltrating | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abbreviated MRI using Dotarem (Experimental): Standard breast MRI studies often have lengthy protocols that make them inherently expensive and time-consuming. Several studies of the use of abbreviated MRI protocols have shown that the shorter protocols have diagnostic accuracy comparable to that of the conventional full MRI protocol. The shorter imaging times achieved with the abbreviated DCE-MRI protocols have the potential to increase efficiency and lower cost by decreasing time in the MRI suite, which in turn may make breast MRI accessible for population-based mass screening. The focus of the proposed research is the investigation of an abbreviated MRI protocol using Dotarem® (Gadoterate Meglumine) by comparing the diagnostic accuracy of dynamic contrast-enhanced breast MRIs performed with an abbreviated protocol versus a full protocol.
  Interventions: Drug: Abbreviated MRI protocol: initial experience with Dotarem® (Gadoterate Meglumine)

INTERVENTIONS:
Drug: Abbreviated MRI protocol: initial experience with Dotarem® (Gadoterate Meglumine) — To test the diagnostic effectiveness of an abbreviated MRI to a full MRI in the evaluation of breast lesions using Dotarem
  Other Names: Abbreviated MRI; Abbreviated MRI with Dotarem; Dotarem

SUMMARY:
Standard breast MRI studies often have lengthy protocols that make them inherently expensive and time-consuming. Several studies of the use of abbreviated MRI protocols have shown that the shorter protocols have diagnostic accuracy comparable to that of the conventional full MRI protocol. There are also promising results of ultrafast DCE-MRI studies with shorter breast MRI protocols that provide not only morphologic but also valuable kinetic information about a lesion. The shorter imaging times achieved with the abbreviated and the ultrafast DCE-MRI protocols have the potential to increase efficiency and lower cost by decreasing time in the MRI suite, which in turn may make breast MRI accessible for population-based mass screening. The focus of the proposed research is the investigation of an abbreviated MRI protocol with ultrafast imaging using Dotarem® (Gadoterate Meglumine).

DETAILED DESCRIPTION:
Breast cancer is second to lung cancer as the leading cause of death among women in the United States. Over 40,000 women were estimated to die of breast cancer in 2016. Early detection is key to improved survival, and overall prognosis is directly linked to the stage of disease at the time of diagnosis. The 5-year relative survival rate has increased since the mid 1970's, in part owing to improvements in early breast cancer detection with screening mammography. Screening with mammography is associated with a 16-40% relative reduction in breast cancer mortality among women aged 40-74 years old, and mammography is the most cost-effective method of breast cancer screening. However, cancers can be missed at mammography, particularly in women with dense breasts. Screening with mammography alone may be insufficient in the screening of women who are at high risk of breast cancer. The need for more effective screening strategies to supplement mammography in these groups of women has led to the use of dynamic contrast-enhanced (DCE) breast MRI. Of the available modalities for evaluation of the breast, MRI has been found to have the highest sensitivity for the detection of breast cancer, irrespective of breast density.

On the basis of evidence from nonrandomized trials and observational studies, breast MRI is indicated as a supplement to mammography for patients at high risk with greater than 20% relative lifetime risk. This cohort of women includes those with: a known BRCA1 or BRCA2 genetic mutation, an approximately 20-25% or greater lifetime risk of breast cancer according to risk assessment tools, a strong family history of beast or ovarian cancer, a history of being treated for Hodgkin's disease and certain genetic syndromes (i.e. Li-Fraumeni syndrome, Cowden syndrome or Bannayan-Riley-Ruvalcaba syndrome). However, for women at intermediate risk, including those with dense breast tissue, screening MRI in the United States is not cost-effective. The cost-effectiveness of screening breast MRI depends on estimated breast cancer incidence and examination cost. The rationale for limiting supplemental screening breast MRI to those at greatest risk is in part due to its high cost.

Investigators have looked at ways of reducing the cost of breast MRI to improve access to it as a supplement screening method for women who are not necessarily in the highest risk group. One way to achieve the efficiency and rapid throughput found with screening mammography is to shorten screening breast MRI protocols, decrease image acquisition time, and shorten image interpretation time. Study results have suggested that shorter protocols and shorter acquisition times can be achieved with maintenance of diagnostic accuracy comparable to that obtained with conventional MRI protocols. Use of these abbreviated MRI protocols could result in lower cost and faster throughput, increasing availability and providing women with dense breasts or at intermediate risk (lifetime risk, 15-20%) greater access to breast MRI.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-80.
* Women with diagnostic imaging findings highly suspicious for breast cancer (BI-RADS category 4 or 5) or known breast cancer (BI-RADS category 6). Per BI-RADS lexicon, category 4 lesions carry a malignancy risk of 2-95% and category 5 lesions carry a malignancy risk of >95%.

Exclusion Criteria:

* Women with a history of adverse reactions to contrast media.
* Women with GFR below 30 mL/min/1.73m².

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Compare the diagnostic accuracy of dynamic contrast-enhanced breast MRIs performed with an abbreviated protocol versus a full protocol | one year
  The abbreviated protocol will be generated from the full diagnostic protocol. It will comprise of a single unenhanced sequence and a single contrast-enhanced sequence. Subtraction images and a maximum intensity projection (MIP) image will be generated post-examination. The novel kinetic information obtained from the early contrast in combination with morphologic information from a high spatial resolution post-contrast scan, may provide unique dynamic parameters to effectively characterize and diagnose breast lesions on MR imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Abe, MD, Principal Investigator — University of Chicago Medicine
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All study details, including study protocol, statistical analysis plan and informed consent plan, will be made available to all researchers through AURA (Automating University-wide Research Administration) -IRB and our electronic medical record.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: the data will be available indefinitely
Access Criteria: Any researcher who wishes to access the data

REFERENCES:
- [Background] Tabar L, Yen MF, Vitak B, Chen HH, Smith RA, Duffy SW. Mammography service screening and mortality in breast cancer patients: 20-year follow-up before and after introduction of screening. Lancet. 2003 Apr 26;361(9367):1405-10. doi: 10.1016/S0140-6736(03)13143-1. PMID 12727392
- [Background] Feig S. Cost-effectiveness of mammography, MRI, and ultrasonography for breast cancer screening. Radiol Clin North Am. 2010 Sep;48(5):879-91. doi: 10.1016/j.rcl.2010.06.002. PMID 20868891
- [Background] Nelson HD, O'Meara ES, Kerlikowske K, Balch S, Miglioretti D. Factors Associated With Rates of False-Positive and False-Negative Results From Digital Mammography Screening: An Analysis of Registry Data. Ann Intern Med. 2016 Feb 16;164(4):226-35. doi: 10.7326/M15-0971. Epub 2016 Jan 12. PMID 26756902
- [Background] Lee CH, Dershaw DD, Kopans D, Evans P, Monsees B, Monticciolo D, Brenner RJ, Bassett L, Berg W, Feig S, Hendrick E, Mendelson E, D'Orsi C, Sickles E, Burhenne LW. Breast cancer screening with imaging: recommendations from the Society of Breast Imaging and the ACR on the use of mammography, breast MRI, breast ultrasound, and other technologies for the detection of clinically occult breast cancer. J Am Coll Radiol. 2010 Jan;7(1):18-27. doi: 10.1016/j.jacr.2009.09.022. PMID 20129267
- [Background] Saslow D, Boetes C, Burke W, Harms S, Leach MO, Lehman CD, Morris E, Pisano E, Schnall M, Sener S, Smith RA, Warner E, Yaffe M, Andrews KS, Russell CA; American Cancer Society Breast Cancer Advisory Group. American Cancer Society guidelines for breast screening with MRI as an adjunct to mammography. CA Cancer J Clin. 2007 Mar-Apr;57(2):75-89. doi: 10.3322/canjclin.57.2.75. PMID 17392385
- [Background] Moore SG, Shenoy PJ, Fanucchi L, Tumeh JW, Flowers CR. Cost-effectiveness of MRI compared to mammography for breast cancer screening in a high risk population. BMC Health Serv Res. 2009 Jan 13;9:9. doi: 10.1186/1472-6963-9-9. PMID 19144138
- [Background] Kuhl CK, Schrading S, Strobel K, Schild HH, Hilgers RD, Bieling HB. Abbreviated breast magnetic resonance imaging (MRI): first postcontrast subtracted images and maximum-intensity projection-a novel approach to breast cancer screening with MRI. J Clin Oncol. 2014 Aug 1;32(22):2304-10. doi: 10.1200/JCO.2013.52.5386. Epub 2014 Jun 23. PMID 24958821
- [Background] Mango VL, Morris EA, David Dershaw D, Abramson A, Fry C, Moskowitz CS, Hughes M, Kaplan J, Jochelson MS. Abbreviated protocol for breast MRI: are multiple sequences needed for cancer detection? Eur J Radiol. 2015 Jan;84(1):65-70. doi: 10.1016/j.ejrad.2014.10.004. Epub 2014 Oct 16. PMID 25454099
- [Background] Harvey SC, Di Carlo PA, Lee B, Obadina E, Sippo D, Mullen L. An Abbreviated Protocol for High-Risk Screening Breast MRI Saves Time and Resources. J Am Coll Radiol. 2016 Apr;13(4):374-80. doi: 10.1016/j.jacr.2015.08.015. Epub 2015 Oct 27. PMID 26521970
- [Background] Tsao J, Kozerke S. MRI temporal acceleration techniques. J Magn Reson Imaging. 2012 Sep;36(3):543-60. doi: 10.1002/jmri.23640. PMID 22903655
- [Background] Kuhl C. The current status of breast MR imaging. Part I. Choice of technique, image interpretation, diagnostic accuracy, and transfer to clinical practice. Radiology. 2007 Aug;244(2):356-78. doi: 10.1148/radiol.2442051620. PMID 17641361
- [Background] Kuhl CK. Current status of breast MR imaging. Part 2. Clinical applications. Radiology. 2007 Sep;244(3):672-91. doi: 10.1148/radiol.2443051661. PMID 17709824
- [Background] Kuhl CK, Schild HH, Morakkabati N. Dynamic bilateral contrast-enhanced MR imaging of the breast: trade-off between spatial and temporal resolution. Radiology. 2005 Sep;236(3):789-800. doi: 10.1148/radiol.2363040811. PMID 16118161
- [Background] Veltman J, Stoutjesdijk M, Mann R, Huisman HJ, Barentsz JO, Blickman JG, Boetes C. Contrast-enhanced magnetic resonance imaging of the breast: the value of pharmacokinetic parameters derived from fast dynamic imaging during initial enhancement in classifying lesions. Eur Radiol. 2008 Jun;18(6):1123-33. doi: 10.1007/s00330-008-0870-8. Epub 2008 Feb 13. PMID 18270714
- [Background] Mann RM, Mus RD, van Zelst J, Geppert C, Karssemeijer N, Platel B. A novel approach to contrast-enhanced breast magnetic resonance imaging for screening: high-resolution ultrafast dynamic imaging. Invest Radiol. 2014 Sep;49(9):579-85. doi: 10.1097/RLI.0000000000000057. PMID 24691143
- [Background] Pineda FD, Medved M, Wang S, Fan X, Schacht DV, Sennett C, Oto A, Newstead GM, Abe H, Karczmar GS. Ultrafast Bilateral DCE-MRI of the Breast with Conventional Fourier Sampling: Preliminary Evaluation of Semi-quantitative Analysis. Acad Radiol. 2016 Sep;23(9):1137-44. doi: 10.1016/j.acra.2016.04.008. Epub 2016 Jun 6. PMID 27283068
- [Background] Abe H, Mori N, Tsuchiya K, Schacht DV, Pineda FD, Jiang Y, Karczmar GS. Kinetic Analysis of Benign and Malignant Breast Lesions With Ultrafast Dynamic Contrast-Enhanced MRI: Comparison With Standard Kinetic Assessment. AJR Am J Roentgenol. 2016 Nov;207(5):1159-1166. doi: 10.2214/AJR.15.15957. Epub 2016 Aug 17. PMID 27532897
- See also: American Cancer Society website. Cancer facts and figures 2016 — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2016.html
- See also: National Cancer Institute website. SEER stat fact sheets:female breast cancer — https://seer.cancer.gov/statfacts/html/breast.html
- See also: American College of Radiology website. ACR Appropriateness Criteria: breast cancer screening. Date of origin 2012. Last review date 2016. — https://acsearch.acr.org/docs/70910/Narrative